CLINICAL TRIAL: NCT00621920
Title: Efficacy Study of Bowel Preparation Before Colonoscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: C.B. Fleet Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PL07.01
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2012-02

CONDITIONS: Bowel Cleansing Prior to Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: FM-601 — Dose-escalation, split dosage, liquid

SUMMARY:
The purpose of this study is to determine the efficacious dose range when used as a bowel preparation before colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Men and nonpregnant women who are scheduled for an elective colonoscopy and who are at least 50 years of age.
* Are able to communicate with study personnel and comply with study requirements.
* Are able and willing to follow study-specified testing, diet, and hydration regimen.
* Have been informed of the nature and risks of the study and have given written informed consent.

Exclusion Criteria:

* Have known or suspected liver disease or any history of abnormal liver function tests.
* Have clinically active cardiovascular disease within the past 6 months.
* Have blood pressure greater than 150/90 mm Hg.
* Have known or suspected renal insufficiency.
* Have known or suspected electrolyte abnormalities, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis, toxic megacolon, or ileus.
* Have a history of prior bowel surgery within 2 years before enrollment, or active inflammatory bowel disease.
* Have diabetes or a history of diabetes.
* Have clinical evidence of dehydration.
* Are pregnant or breast-feeding.
* Are unwilling to abstain from alcohol consumption from one day before colonoscopy until discharged from the study.
* Use prohibited medications of the study in the defined timeframes.
* Have received any investigational agent within 30 days before dosing.
* Have any known contraindications to the study treatment.
* Have any known or suspected allergies to the components of the study medication.
* Have any other condition which would make the subject unsuitable for inclusion in the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Effectiveness of bowel cleansing based on a grading scale. | During colonoscopy

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Advanced Clinical Research Institute, Anaheim, California
  - Qualia Clinical Services, Omaha, Nebraska